CLINICAL TRIAL: NCT05252455
Title: A Randomized Controlled Trial to Evaluate the Effects of Pelvic and Abdominal Mechanical Exercises During Pregnancy on Reducing the Rate of Cesarean Section and Preventing Pelvic Floor Dysfunction Diseases
Brief Title: A RCT to Evaluate the Effects of Pelvic and Abdominal Mechanical Exercises During Pregnancy on Reducing the Rate of CS and Preventing PFD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qiu Jin (Other)
Responsible Party: Sponsor-Investigator, Qiu Jin, Executive director of Obstetrics and Gynecology, Shanghai Tong Ren Hospital
Organization: Shanghai Tong Ren Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prof. Qiu Jin
Record Dates: First submitted 2021-12-25; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Mode of Delivery; Pelvic Floor Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Other): pelvic and abdominal mechanics exercise
  Interventions: Behavioral: pelvic and abdominal mechanics exercise
- control group (No Intervention): Normal prenatal examination

INTERVENTIONS:
Behavioral: pelvic and abdominal mechanics exercise — starting from 24 weeks of pregnancy, participate in the pelvic and abdominal mechanics exercises offered by the "Good Pregnancy" College of Shanghai Tongren Hospital once a week. Each class lasts one hour until the 38th week of pregnancy (attend at least 10 times)
  Arms: exercise group

SUMMARY:
Pelvic floor dysfunction diseases seriously affect the quality of life. Childbirth, especially vaginal birth, is significantly related to pelvic floor dysfunction diseases, which mainly cause urinary incontinence and pelvic organ prolapse. Studies have found that exercise during pregnancy can help reduce the rate of caesarean section and prevent the occurrence of organic pelvic floor disorders. Pregnant women without obvious comorbidities should be encouraged to participate in fitness programs that include core muscle exercises.

At present, there is no clinical research data about the influence of pelvic and abdominal mechanical exercise during pregnancy on the way of delivery and postpartum pelvic floor rehabilitation.

This study is a clinical randomized controlled study, use pelvic and abdominal mechanical exercises during pregnancy to train proprioception of the pelvis, increase local muscle strength, ensure physical strength while taking into account flexibility, to evaluate the impact of pelvic and abdominal mechanical exercises during pregnancy on the cesarean section rate of primiparas and on Prevention of pregnancy-related pain during pregnancy and postpartum pelvic floor dysfunction diseases.To provide strong evidence-based medical evidence for the promotion of pelvic and abdominal mechanical exercise during pregnancy in the majority of pregnant women in the future.

DETAILED DESCRIPTION:
This study is a clinical randomized controlled study, which aims to evaluate the influence of pelvic and abdominal mechanical exercise during pregnancy on pregnancy outcome and pelvic floor health, and to provide strong evidence-based medical evidence for the promotion of pelvic and abdominal mechanical exercise during pregnancy in the majority of pregnant women in the future.

Pregnant women included in the study must be pregnant women who gave birth during the formal examination in the Obstetrics Department of Shanghai Tongren Hospital during the study period and met the enrollment criteria.

The researchers randomly divided pregnant women into two groups: exercise group and control group. The sports group or control group cards are printed and placed in an opaque envelope, which will be stored and locked in the cabinet. The recruited pregnant women select an envelope from the available envelopes to determine the group selection, and plan to enroll 10 cases each month.

Pregnant women in the exercise group will participate in the pelvic and abdominal mechanics exercise course offered by Tongren Hospital's Obstetrics Department once a week from the 24th week of pregnancy to the 38th week. The professionally certified Li Yueyue will be the coach. During this period, the pregnant women in the control group will receive the same formal prenatal examinations Maternity school curriculum (including Lamez breathing method, nutrition and weight management guidance during pregnancy, etc.), a comparative analysis of relevant evaluation indicators during pregnancy, delivery and 42-day follow-up results after delivery.

ELIGIBILITY:
Inclusion Criteria:

1. The primipara who is 18 years old ≤ the age at delivery ≤ 38 years old (this pregnancy is the pregnant woman who gave birth for the first time);
2. Singleton pregnancy;
3. 22-24 weeks of pregnancy;
4. Pregnant women voluntarily signed an informed consent form to participate in this study.

Exclusion Criteria:

1. Cervical insufficiency;
2. People with low placenta (the lower edge of the placenta is less than 2 cm from the inner cervical opening);
3. Severe medical and surgical diseases before pregnancy (such as hypertension, cardiac insufficiency, arrhythmia, etc.);
4. Twin and multiple pregnancy;
5. Mid-Tang, non-invasive DNA or large row malformations suggest fetal malformations;
6. Pregnant women have genital malformations (vaginal diaphragm, uterine malformations, etc.);
7. Those who plan to participate in regular aerobic exercises during pregnancy.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | 2 years
  Cesarean section rate for pregnant women who give birth at 37 weeks of gestation and later (full-term)

SECONDARY OUTCOMES:
Pelvic floor dysfunction | 2 years
  Pelvic floor impact questionnaire-short form 7 (PFIQ-7). This questionnaire score scale is 0-100, higher scores mean a worse outcome.1-32 means minor distress,33-66 means moderate distress,67-100 means severe distress.

CONTACTS AND LOCATIONS:
Overall Officials: jin Qiu, Principal Investigator — Shanghai Tongren Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appropriate technology for birth. Lancet. 1985 Aug 24;2(8452):436-7. PMID 2863457
- [Background] Lumbiganon P, Laopaiboon M, Gulmezoglu AM, Souza JP, Taneepanichskul S, Ruyan P, Attygalle DE, Shrestha N, Mori R, Nguyen DH, Hoang TB, Rathavy T, Chuyun K, Cheang K, Festin M, Udomprasertgul V, Germar MJ, Yanqiu G, Roy M, Carroli G, Ba-Thike K, Filatova E, Villar J; World Health Organization Global Survey on Maternal and Perinatal Health Research Group. Method of delivery and pregnancy outcomes in Asia: the WHO global survey on maternal and perinatal health 2007-08. Lancet. 2010 Feb 6;375(9713):490-9. doi: 10.1016/S0140-6736(09)61870-5. Epub 2010 Jan 11. PMID 20071021
- [Background] Qiao J, Wang Y, Li X, Jiang F, Zhang Y, Ma J, Song Y, Ma J, Fu W, Pang R, Zhu Z, Zhang J, Qian X, Wang L, Wu J, Chang HM, Leung PCK, Mao M, Ma D, Guo Y, Qiu J, Liu L, Wang H, Norman RJ, Lawn J, Black RE, Ronsmans C, Patton G, Zhu J, Song L, Hesketh T. A Lancet Commission on 70 years of women's reproductive, maternal, newborn, child, and adolescent health in China. Lancet. 2021 Jun 26;397(10293):2497-2536. doi: 10.1016/S0140-6736(20)32708-2. Epub 2021 May 24. No abstract available. PMID 34043953
- [Background] Bacchi M, Mottola MF, Perales M, Refoyo I, Barakat R. Aquatic Activities During Pregnancy Prevent Excessive Maternal Weight Gain and Preserve Birth Weight: A Randomized Clinical Trial. Am J Health Promot. 2018 Mar;32(3):729-735. doi: 10.1177/0890117117697520. Epub 2017 Mar 9. PMID 28279085